CLINICAL TRIAL: NCT02634736
Title: A Multi-centre, Cluster Randomised Controlled Trial Comparing Falls Prevention Exergames With Remote Monitoring Against Standard Falls Prevention Programmes for Community Dwelling Older Adults at Risk of Falls.
Brief Title: Cluster RCT of Falls Prevention Exergames for Older Adults
Acronym: Profexs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Dr Emma Stanmore, Dr, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R119047/195378
Record Dates: First submitted 2015-12-09; First posted 2015-12-18 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Accidental Falls

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exergame plus usual treatment (Experimental): Exergame programme plus usual falls prevention treatment including assessment and exercises (prescribed by the physiotherapists).
  Interventions: Device: Exergame plus usual treatment
- Usual treatment (No Intervention): No exergame programme, just usual falls prevention treatment including assessment and exercises (prescribed by the physiotherapists).

INTERVENTIONS:
Device: Exergame plus usual treatment — An individualised [i.e. frequency and duration will be set according to each participant's baseline levels] Exergame programme incorporated into participant's normal routines plus usual falls prevention treatment (prescribed by the physiotherapists).
  Arms: Exergame plus usual treatment

SUMMARY:
This cluster RCT study will investigate the effectiveness of strength/balance Exergames (exercise and computer games that use body movements as controls) developed to improve balance, function, prevent falls and increase exercise adherence for older people in the home setting. The proposal incorporates postural stability Exergames that have been developed with users based on best evidence strength and balance exercise (OTAGO and Postural Stability) currently used by therapists, safe for older people and can be used in the home setting

DETAILED DESCRIPTION:
STUDY OBJECTIVES

Primary Question:

To determine the effect of using MIRA falls prevention Exergames to improve balance in older adults.

Secondary Question/Objectives:

1. What features of usual falls prevention teams routines/activities need consideration for successful implementation of the strength and balance Exergame intervention?
2. How can the Exergames be tailored for home use for older adults?
3. What are the most effective outcome measurements to detect meaningful changes resulting from the MIRA Exergame programme?
4. What are the current challenges and solutions to accessing robust data depicting costs of current therapy treatment compared to home-based MIRA Exergame treatment?
5. Is it possible to retain participants in the intervention during the 12-week MIRA Exergame intervention with respect to outcomes including motivation, enjoyment and usability?
6. What training and support needs are required to maximise the use of the MIRA Exergame technology?
7. What are the costs of the MIRA Exergame intervention and how cost-effectiveness is the MIRA Exergame intervention compared with usual care.
8. What are the effects on falls and fall-related use of health services during a 6-month follow up? STUDY DESIGN & PROTOCOL Participants This project is a cluster RCT study to test the effectiveness of undertaking MIRA Exergames in the sheltered home setting in addition to usual activities. A maximum of 12 sheltered housing units, with 108 participants will be recruited to participate in the study. These will be split into the experimental group (6 sheltered housing units with n=54) and the control group (6 sheltered housing units with n=54). These 2 groups will be based in 2 falls prevention teams in Manchester and a second site in Glasgow.

Falls prevention team staff and other professionals will also be recruited into the study (n=20) to either give their professional insights and feedback on the usability of the exergames and/or help supervise the participants.

Study Intervention Sheltered Housing facilities will be recruited via the Manchester and Glasgow Housing Associations to enable facilities of similar size and deprivation status to be identified. The sheltered housing facilities will be randomised into two groups: the Exergame/experimental group (n=6 sheltered housing units with 9 participants recruited in each); and the control group (n=6 sheltered housing units with 9 participants recruited in each). The participants in the control groups will be offered the Exergame intervention after the final 12-week measurements for ethical reasons. A pre-enrolment examination will be carried out by a trained research physiotherapist to assess each person's suitability to participate in the Kinect exergame programme, and also evaluate potential impact of the Exergames on various aspects of their physical health. Their GPs will also be notified.

The eligible participants will be given a tailored, individualised [i.e. frequency and duration will be set according to each participant's baseline levels] Exergame programme incorporated into their normal routines plus usual falls prevention treatment (prescribed by the physiotherapists). The control group will be given usual falls prevention assessment, treatment and home exercises without the Exergames. The Exergame intervention will run for 12 weeks to test the efficacy of the intervention. Outcome measures to be used during these 12 weeks will include a series of standardised tests and questionnaires. Each participant will be aided in completing these measures. These assessments will take place 3 times: at baseline, 6 weeks, and at the end of the 12-week period.

The intervention participants will be offered the use the Exergame intervention in a group setting and/or home setting according to their preferences (previously piloted in a small feasibility study). The physiotherapists and physiotherapist assistants will supervise and monitor their progress and will also have the ability to see the results of the Exergame programme (anonymised data on points gained, time used, range of motion) at the Falls Prevention Clinic for participants that consent to the sharing of this anonymised data.

At the end of the 12 weeks, focus groups and interviews will be conducted to assess the therapists and participants' perspectives regarding the effectiveness of the remote MIRA Exergame programmes and their usability.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for recruiting participants:

1. able to use gaming technology safely as assessed by the therapist, with access to television and a 2m space in the home to exercise safely (Note: Kinect-based Exergame system does not require the use of any hand-held consoles; and the exercises will be customised/tailored to each participant's needs, including those having difficulty standing a long time);
2. participants will be home-dwelling participants aged 60 years and above;
3. participants should be able to watch TV with or without glasses from a 2m distance;
4. participants should be English-speaking, and registered with primary care general practices; and
5. participants must have the mental capacity to give informed consent.

Exclusion Criteria:

1. currently using gaming technologies to exercise;
2. inability to comprehend the study procedures;
3. acute illness, severe congestive cardiac failure, uncontrolled hypertension, recent fracture or surgery;
4. Myocardial Infarction or Stroke in past 6 months;
5. severe cognitive impairment;
6. orthopaedic surgery in last 6 months, or on waiting list to have orthopaedic surgery;
7. wheelchair users;
8. severe auditory or visual impairment; and
9. peripheral neuropathy or other uncontrolled medical conditions likely to compromise the ability to exercise.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2016-02; Primary Completion 2017-02 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Balance | 12 weeks
  The Berg Balance Scale (BBS)

SECONDARY OUTCOMES:
Adherence | 12 weeks
  Duration in minutes of use of the Exergames
Physical activity levels | 12 weeks
  The Physical Activity Scale for the Elderly to assess user's physical activity levels
Lower limb strength | 12 weeks
  Timed up and go measurement of lower limb strength
Fear of falling | 12 weeks
  The Short Falls Efficacy Scale-International (FES-I) The FES-I is a validated and reliable 7-item tool that measures confidence in performing a range of activities of daily living without falling
Cognition | 12 weeks
  The Addenbrooke's Cognitive Examination III (ACEIII) to measure cognition levels in older adults
Mood | 12 weeks
  The 5-item Geriatric Depression Scale screening tool for depression in older adults

CONTACTS AND LOCATIONS:
Overall Officials: Emma K Stanmore, PhD, Principal Investigator — University of Manchester
Locations (1):
- Dr Emma Stanmore, Manchester, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stanmore EK, Mavroeidi A, de Jong LD, Skelton DA, Sutton CJ, Benedetto V, Munford LA, Meekes W, Bell V, Todd C. The effectiveness and cost-effectiveness of strength and balance Exergames to reduce falls risk for people aged 55 years and older in UK assisted living facilities: a multi-centre, cluster randomised controlled trial. BMC Med. 2019 Feb 28;17(1):49. doi: 10.1186/s12916-019-1278-9. PMID 30813926